CLINICAL TRIAL: NCT06313827
Title: Effectiveness of an e-Health Program to Prevent Exacerbations in the Cystic Fibrosis Population: a Randomized Clinical Trial
Brief Title: e-Health Program to Prevent Exacerbations in the Cystic Fibrosis Population
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: Asociación de Fibrosis Quística - Comunidad Valenciana (Unknown)
Responsible Party: Principal Investigator, SARA CORTES AMADOR, Assistant lecturer PhD in Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: UV-INV_3165929
Record Dates: First submitted 2024-03-01; First posted 2024-03-15 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cystic Fibrosis
Keywords: e-Health; physiotherapy; Cystic fibrosis; exacerbation; quality of life
MeSH Terms: conditions — Cystic Fibrosis | interventions — Exercise; KTN1 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be randomly assigned to one of three study groups by the person conducting the intervention.
  All participants receive usual physiotherapy treatment, and both intervention groups receive monitoring and follow-up of their clinical situation.
  The evaluators are unaware of the assignment at all times.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control exercise group (CG-1) (Active Comparator): Participants will receive their usual physiotherapy treatment.
  Interventions: Behavioral: Exercise Group (CG-1)
- Exercise plus monitoring group (TG-2) (Experimental): Participants will receive their usual physiotherapy treatment, plus explanation of the use of the monitoring equipment.
  Interventions: Behavioral: Exercise plus Monitoring Group (TG-2)
- Exercise plus monitoring and follow-up group (TGF-3) (Experimental): Participants will receive their usual physiotherapy treatment, plus explanation of the use of the monitoring equipment, plus telematic control (via 1:1 real-time videoconferencing) of exacerbations with feedback from the physiotherapist.
  Interventions: Behavioral: Exercise plus monitoring and follow-up group (TGF-3)

INTERVENTIONS:
Behavioral: Exercise plus Monitoring Group (TG-2) — Participants will receive their usual physiotherapy treatment and user education on bronchial care and hygiene, plus a dossier on the use of monitoring equipment such as: pulse oximeter, thermometer, digital spirometer, Medical Research Council dyspnoea scale. If the patient detects an exacerbation (due to symptoms or monitoring of the equipment), they can contact a physiotherapist who can adjust the treatment.
  Other Names: Exercise plus Monitoring Group
  Arms: Exercise plus monitoring group (TG-2)
Behavioral: Exercise plus monitoring and follow-up group (TGF-3) — Participants who will receive their usual physiotherapy treatment and user education on bronchial care and hygiene, plus dossiers on the use of monitoring equipment ; plus telematic control of exacerbations (questionnaires and monitoring of the parameters of the aforementioned equipment). Depending on the follow-up, physiotherapy treatment will be adjusted.
  The questionnaire includes tracking of the following parameters: cough, secretions (quantity, colour, viscosity), chest tightness, dyspnoea, exercise tolerance, tiredness and appetite).
  The follow-up will consist of weekly filling the spreadsheet to which the physiotherapist will have access and who, by reviewing the parameters, will be able to adjust the treatment. The physiotherapist will systematically make videocalls to the participants and if the follow-up values require it, he/she will call every week.
  Arms: Exercise plus monitoring and follow-up group (TGF-3)
Behavioral: Exercise Group (CG-1) — Participants who will receive their usual physiotherapy treatment and user education on bronchial care and hygiene
  Other Names: Exercise Group
  Arms: Control exercise group (CG-1)

SUMMARY:
The goal of this clinical trial is to analyse the impact of a telematic assessment and monitoring protocol in people with cystic fibrosis, in order to identify exacerbations early, thus preventing loss of lung function and maintaining quality of life.

Participants will be assigned to one of 3 study groups:

Control group (CG-1): will receive their usual physiotherapy treatment; Treatment group (TG-2): will receive their usual physiotherapy treatment, plus explanation of the use of the monitoring equipment; Treatment and follow-up group (TGF-3): will receive their usual physiotherapy treatment, plus explanation of the use of the monitoring equipment, plus telematic control of exacerbations with feedback from the physiotherapist.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cystic fibrosis
* Family access to an internet-enabled device
* Camera and microphone
* Absence of exacerbations in the last 30 days

Exclusion Criteria:

* Patients with lung transplant or on the waiting list for lung transplantation
* Previous eye surgery (3 months)
* Hemothorax
* Active infection or inflammatory process
* Tumors
* Cognitive problems that make it impossible for them to use telematic devices.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Clinical exacerbation | At baseline (T1), at 6 months (T2) and at 12 months(T3).
  Presence of an exacerbation. To consider this the Escribano criteria will be followed, for which the presence of at least 3 of the criteria stablished (Clinical, spirometric, radiographic, analytical, and microbiological), collected by interviewing the patient

SECONDARY OUTCOMES:
Dyspnea | At baseline (T1), at 6 months (T2) and at 12 months(T3).
  Modified Medical Research Council (mMRC) scale (0 to 4 points). Higher scores are related to higher dyspnea.
Spirometric function | At baseline (T1), at 6 months (T2) and at 12 months(T3).
  Forced expiratory volume in the first second (FEV1) in L/sec
Oxigenation | At baseline (T1), at 6 months (T2) and at 12 months(T3).
  Oxyhemoglobin saturation in percent.
Functional capacity | At baseline (T1), at 6 months (T2) and at 12 months(T3).
  30 seconds sit-to-stand test (in number of repetitions)
Quality of life (QoL) | At baseline (T1) and at 12 months(T3).
  Cystic fibrosis questionnaire-revised (in score points). It is a 0-100 scale with higher scores indicating better quality of life.

OTHER OUTCOMES:
Motivation to engage in physical activity | At baseline (T1)
  A confidential online ad-hoc 13-item survey regarding their views, opinions and practices in relation to physical activity. This is a survey that is analyzed qualitatively.

CONTACTS AND LOCATIONS:
Locations (1):
- Instalaciones de la Universitat de Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No